CLINICAL TRIAL: NCT03087344
Title: Postprandial Liver and Spleen Stiffness Measurements in the Noninvasive Diagnosis of Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0042
Record Dates: First submitted 2017-03-06; First posted 2017-03-22 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Chronic Liver Disease
Keywords: Postprandial liver and spleen stiffness measurements; Transient elastography; Cirrhosis; Acoustic radiation force impulse
MeSH Terms: conditions — Fibrosis | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Intervention Model Description: Cross sectional diagnostic study of Chronic liver disease patients who have had a liver stiffness measurement performed that is discordant with clinical impression either clinically the patient appears to have cirrhosis but liver stiffness measurement is less than 10 kPa or clinically there is no evidence of cirrhosis but there liver stiffness measurement is more than 15 kPa or the patients liver stiffness measurement is in the grey zone which means patients' liver stiffness measurement is between 10 and 15 kPa to investigate the utility of postprandial postprandial liver and spleen stiffness measurements in the noninvasive diagnosis of cirrhosis
Masking Description: All the above, the patient, provider and investigator and outcome assessor will not know the result of the biopsy to know if the participant does or does not have cirrhosis at the time of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Chronic liver disease (Experimental): patient who will undergo liver biopsy will undergo liver stiffness and spleen stiffness will be measured before and after a standard meal is administered by Fibroscan and Acoustic Radiation Force Impulse
  Interventions: Device: Fibroscan and Acoustic Radiation Force Impulse; Device: Fibroscan; Device: Acoustic Radiation Force Impulse

INTERVENTIONS:
Device: Fibroscan and Acoustic Radiation Force Impulse — Liver stiffness and spleen stiffness will be measured before and after a standard meal is administered by Fibroscan and Acoustic Radiation Force Impulse
Device: Fibroscan — Liver stiffness will be measured before and after a standard meal is administered
  Other Names: Transient elastography
Device: Acoustic Radiation Force Impulse — Liver stiffness and spleen stiffness will be measured before and after a standard meal is administered by Fibroscan and Acoustic Radiation Force Impulse

SUMMARY:
This is a study that will evaluate the utility of measuring liver and spleen stiffness before and after a meal by a non invasive ultrasound based technologies called Fibroscan (Transient elastography) and acoustic radio-frequency impulse (ARFI) in diagnosing or excluding cirrhosis in patients with chronic liver disease who will be getting a liver biopsy.

DETAILED DESCRIPTION:
This is a prospective longitudinal study that will evaluate the utility of change in liver stiffness (LSM) and spleen stiffness measurements after a test meal in patients whom the diagnosis cannot be reliably ruled in or ruled out based on two measurement of LSM by TE per standard of care. This includes patients in whom there is discordance between clinical impression and LSM and/or LSM are in the grey zone (LSM between 10 and 15 kPa). Liver biopsy/HVPG which is performed as standard of care will be used as gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85
* History of chronic liver disease who have had a liver stiffness measurement performed that is discordant with clinical impression (clinically the patient appears to have cirrhosis but LSM <10) or clinically there is no evidence of cirrhosis but LSM>15) or LSM are in the grey zone (LSM between 10 and 15 kPa)

Exclusion Criteria:

* Any signs of decompensated cirrhosis (e.g., jaundice, ascites, variceal hemorrhage, or hepatic encephalopathy)
* Hepatocellular carcinoma
* Patients with chronic Hep C who have undergone antiviral therapy
* Ongoing alcohol abuse
* Acute hepatitis
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in liver and spleen stiffness from pre and post meal obtained by Fibroscan | 30 minutes interval between the two measurements of liver stiffness from pre meal to post meal
  Liver stiffness will be obtained by fibroscan in kPa, Liver stiffness will be obtained pre and post meal, the delta change of liver stiffness will be computed in an AUROC to see the Sensitivity, specificity, positive predictive value and negative predictive value of the delta change and diagnosing or excluding cirrhosis

SECONDARY OUTCOMES:
Change in liver and spleen stiffness from pre and post meal obtained by ARFI | 30 minutes interval between the two measurements of liver and spleen stiffness from pre meal to post meal
  Liver and spleen stiffness will be obtained by ARFI in m/sec, Liver and spleen stiffness will be obtained pre and post meal, the delta change of liver and spleen stiffness will be computed in an AUROC to see the Sensitivity, specificity, positive predictive value and negative predictive value of the delta change and diagnosing or excluding cirrhosis

CONTACTS AND LOCATIONS:
Overall Officials: Guadalupe Garcia-Tsao, MD, Principal Investigator — Yale and VA
Locations (1):
- Wesy haven va, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided
once all data is collected, possibly share individual data